CLINICAL TRIAL: NCT00673634
Title: Efficiency of Preoxygenation in Obese Patients: Evaluation of Traditional Method Versus Pressure Assisted Preoxygenation.
Brief Title: Efficiency of Preoxygenation in Obese Patients: Pressure Assisted Versus Traditional Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Mihai Georgescu / anesthesiology resident, Maisonneuve-Rosemont Hospital / Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 07122
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
Keywords: preoxygenation; method; efficiency; obesity; BiPAP; FeO2
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard preoxygenation
  Interventions: Procedure: Standard preoxygenation
- 2 (Active Comparator): BiPAP assisted preoxygenation
  Interventions: Procedure: BiPAP assisted preoxygenation

INTERVENTIONS:
Procedure: Standard preoxygenation — Spontaneous breathing of 100% oxygen in a facemask for 3 minutes.
  Arms: 1
Procedure: BiPAP assisted preoxygenation — Spontaneous breathing of 100% oxygen in a facemask with application of an inspiratory pressure of 4cm H2O and a positive end-expiratory pressure of 4cm H2O, for 3 minutes.
  Arms: 2

SUMMARY:
The purpose of this clinical trial is to evaluate whether pre-oxygenation of obese patients with BiPAP 4cm H2O, renders any benefit to the quality of pre-oxygenation measured by the expired oxygen fraction (FeO2) and whether it is as well tolerated as the traditional method of spontaneous breathing for 3 minutes.

DETAILED DESCRIPTION:
Traditional pre-oxygenation in obese patients has been proven to allow a time of apnea far reduced when compared with patients closer to their ideal body weight. This effect is attributable to several factors :

* Reduced FRC
* Increased closing capacity
* Diminished tidal volume due to increased resistance of the airway, diminished compliance of the thoracic cage and diminished strength and endurance of respiratory muscles.
* Increase in atelectasis formation upon induction of general anaesthesia.
* Increased O2 consumption due to the increased workload of respiratory muscles and to the general increase in metabolism.
* Increase in true shunt. Studies have demonstrated a reduction in atelectasis formation by application of CPAP during pre-oxygenation and PEEP during anaesthesia. Also, 25º inclination of the patient in the supine position, on the operating table, has demonstrated prolongation of time of apnea in a significant amount. Outside the operating room, PEEP of 5 cmH2O has been demonstrated useful in prolonging time of apnea when used during pre-oxygenation in hypoxic patients requiring tracheal intubation in the intensive care.

Yet, few studies have evaluated BiPAP in the operating room setting as to the effect on FeO2 and to the tolerance by the patients.

Thus, it is our intent to evaluate the efficiency of application of an inspiratory assistance pressure of 4cmH2O and PEEP 4cmH2O during a 3 minutes pre-oxygenation trial as to the level of FeO2 attained, the rate of attainment of FeO2 > 90% and the tolerance by the patient of the procedure, when compared with a 3 minute trial of the traditional method.

For this purpose, consenting, non pre-medicated obese patients scheduled for surgery in the operating ward of our institution will be brought earlier to the operating room, the day of their surgery. In an idle operating room, they will go through two trials of 100% O2 pre-oxygenation lasting 3 minutes each, at an interval of 20 minutes during which the patients will rest in a semi-sitting position, breathing spontaneously at ambient air. The order of the two trials will be randomly assigned between standard pre-oxygenation vs BiPAP pre-oxygenation. Both patients and anesthesia assistants providing the pre-oxygenation will be blinded as to the ongoing trial. Data from the anesthesia machine will be recorded visually to be analysed subsequently by a blinded third party. During each trial, the comfort of the patient on a local 4 point scale will be graded every minute.

At the end of the study period, patients will be returned to the waiting area of the operating ward before the scheduled time of their surgery. The protocol is intended to not interfere with the planned anesthesia technique or the surgery in any way.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Scheduled for surgery

Exclusion Criteria:

* Non fasted patient
* Clinically significant gastro-oesophageal reflux
* Intestinal occlusion
* Presence of nasogastric tube
* Facial hair
* Claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
rate of increase of fractional expired oxygen level | every 10 seconds during each 3 minute preoxygenation period

SECONDARY OUTCOMES:
Level of fractional expired oxygen. Patient tolerance. Ease of preoxygenation administration. Presence of secondary effects (gastric reflux, respiratory discomfort, burps) | every minute during each 3 minute preoxygenation trial and at the end of each trial

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Drolet, MD, FRCPC, Study Director — Maisonneuve-Rosemont Hospital; Mihai L Georgescu, MD, resident, Principal Investigator — Maisonneuve-Rosemont Hospital / Université de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] HAMILTON WK, EASTWOOD DW. A study of denitrogenation with some inhalation anesthetic systems. Anesthesiology. 1955 Nov;16(6):861-7. doi: 10.1097/00000542-195511000-00004. No abstract available. PMID 13268902
- [Background] Campbell IT, Beatty PC. Monitoring preoxygenation. Br J Anaesth. 1994 Jan;72(1):3-4. doi: 10.1093/bja/72.1.3. No abstract available. PMID 8110546
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Wax DB. Mechanism of benefit of head-up preoxygenation in obese patients. Anesthesiology. 2006 Feb;104(2):381; author reply 381. doi: 10.1097/00000542-200602000-00035. No abstract available. PMID 16436870
- [Background] Pelosi P, Ravagnan I, Giurati G, Panigada M, Bottino N, Tredici S, Eccher G, Gattinoni L. Positive end-expiratory pressure improves respiratory function in obese but not in normal subjects during anesthesia and paralysis. Anesthesiology. 1999 Nov;91(5):1221-31. doi: 10.1097/00000542-199911000-00011. PMID 10551570
- [Background] Parameswaran K, Todd DC, Soth M. Altered respiratory physiology in obesity. Can Respir J. 2006 May-Jun;13(4):203-10. doi: 10.1155/2006/834786. PMID 16779465
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Goldberg ME, Norris MC, Larijani GE, Marr AT, Seltzer JL. Preoxygenation in the morbidly obese: a comparison of two techniques. Anesth Analg. 1989 Apr;68(4):520-2. No abstract available. PMID 2494907
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Background] Rose DK, Cohen MM. The airway: problems and predictions in 18,500 patients. Can J Anaesth. 1994 May;41(5 Pt 1):372-83. doi: 10.1007/BF03009858. PMID 8055603
- [Background] Gagnon C, Fortier LP, Donati F. When a leak is unavoidable, preoxygenation is equally ineffective with vital capacity or tidal volume breathing. Can J Anaesth. 2006 Jan;53(1):86-91. doi: 10.1007/BF03021532. PMID 16371614
- [Background] Ho-Tai LM, Devitt JH, Noel AG, O'Donnell MP. Gas leak and gastric insufflation during controlled ventilation: face mask versus laryngeal mask airway. Can J Anaesth. 1998 Mar;45(3):206-11. doi: 10.1007/BF03012903. PMID 9579256
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] Berthoud MC, Peacock JE, Reilly CS. Effectiveness of preoxygenation in morbidly obese patients. Br J Anaesth. 1991 Oct;67(4):464-6. doi: 10.1093/bja/67.4.464. PMID 1931404
- [Background] Kashyap L, Yaddanapudi LN, Sandhya. Arterial desaturation during induction with and without preoxygenation: evaluation of four techniques. Anaesth Intensive Care. 1993 Dec;21(6):811-3. doi: 10.1177/0310057X9302100611. PMID 8122739
- [Background] Rapaport S, Joannes-Boyau O, Bazin R, Janvier G. [Comparison of eight deep breaths and tidal volume breathing preoxygenation techniques in morbid obese patients]. Ann Fr Anesth Reanim. 2004 Dec;23(12):1155-9. doi: 10.1016/j.annfar.2004.10.012. French. PMID 15589355